CLINICAL TRIAL: NCT05521893
Title: Effectiveness of Telemedicine Care Replacing Standard Care in Gestational Diabetes: a Randomized Controlled Trial
Brief Title: Effectiveness of Telemedicine Care Replacing Standard Care in Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-302/2020-4
Record Dates: First submitted 2022-06-27; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-06

CONDITIONS: Gestational Diabetes
Keywords: telemedicine; glycemic control; perinatal outcomes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine group (Experimental)
  Interventions: Other: Telemedicine care
- Standard care group (Active Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Telemedicine care — In the telemedicine group, the appointments are performed online via scheduled videoconferences, on a monthly basis.
  All women in the telemedicine group receive a smartphone with the installed application that enable transfer of the measured capillary glucose concentration.
  Arms: Telemedicine group
Other: Standard care — In the standard care group, visits are scheduled at the diabetes clinic on a monthly basis.
  Arms: Standard care group

SUMMARY:
This is a a single-centre, parallel, randomized controlled trial in women with gestational diabetes mellitus (GDM). Women are randomized to routine monthly prenatal clinic care (standard care group) or a group sending daily glucose readings via an application installed on a smartphone and monthly individual videoconferences replacing in-person visits (telemedicine group). The overall aim is to compare the effectiveness of the combine synchronous and asynchronous telemedicine care with the standard care in women with GDM.

DETAILED DESCRIPTION:
In our single-centre, parallel, randomized controlled trial in women with gestational diabetes (GDM) the investigators aim to compare the effectiveness of combined synchonous and asynchronous telemedicine care with the standard care.

In the telemedicine group appointments are performed online via monthly scheduled videoconferences. Women also receive a smartphone with the installed application that enable transfer of the measured capillary glucose concetration at the same time it is performed. The glucose data sent by women are reviewed once per week and after that healthcare professionals contact women if necessary. On the other hand, in the standard care group, visits are scheduled normally on a monthly basis at the diabetes clinic.

Intention-to-treat analysis is going to be performed. The investigators aim to compare glycemic control, gestational weight gain and perinatal data between groups.

Student's t-test or Mann-Whitney U test will be used for normally or non-normally distributed variables. Differences between groups in categorical data will be calcuated by Chi square.

ELIGIBILITY:
Inclusion Criteria:

* less then 30 weeks of gestation at enrolement
* GDM diagnosis
* at least moderate Slovenian language skills
* willingness to participate

Exclusion Criteria:

* more than 30 weeks of pregnancy
* overt diabetes or fasting glucose >6.9 mmol/l at diagnosis
* multiple pregnancy
* poor Slovene language skills
* history or bariatric surgery or other surgeries that induce malabsorbtion
* use of systemic steroids prior to enrolment
* presence of concomitant disease that could affect glucose control or self-management (e.g. uncontrolled psychiatric disorder)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Average fasting glucose concentration | 1 month
  Average fasting based on participant's SMBG in the 3rd trimester
Percentage of glucose readings in the target range | 1 month
  average percentage for the 3rd trimester
Compliance with SMBG | 1 month
  is defined as defined as the number of actual glucose measurements performed divided by the number of recommended glucose measurements*100
The percentage of individuals needing insulin treatment | once during pregnancy
Average postprandial glucose concentration | 1 month
  Average postprandial glucose based on participant's SMBG in the 3rd trimester

SECONDARY OUTCOMES:
gestational weight gain | once during pregnancy
  from pre-conception until labour
Newborn birth weight | delivery
LGA incidence | delivery
Gestational age at birth | delivery
Preterm birth | delivery
Incidence of preeclampsia | delivery
Incidence of caesarean section | delivery

CONTACTS AND LOCATIONS:
Overall Officials: Drazenka Pongrac Barlovic, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Munda A, Mlinaric Z, Jakin PA, Lunder M, Pongrac Barlovic D. Effectiveness of a comprehensive telemedicine intervention replacing standard care in gestational diabetes: a randomized controlled trial. Acta Diabetol. 2023 Aug;60(8):1037-1044. doi: 10.1007/s00592-023-02099-8. Epub 2023 Apr 25. PMID 37185903